CLINICAL TRIAL: NCT04226599
Title: Evaluation of the Safety and Efficacy of the Peripheral Scoring Drug Balloon (Dissolve AV) in Treatment of Hemodialysis Arteriovenous Fistulae Stenosis A Prospective Multicenter Randomized Controlled Clinical Study
Brief Title: A Safety and Efficacy Study of Hemodialysis Arteriovenous Fistulae Stenosis Treated With DissolveAV
Acronym: DissolveAVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DK Medical Technology (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VP-P-2018-018
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Fistulas Arteriovenous
Keywords: Dialysis scoring Fistulas
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dissolve AVF Group (Experimental): This group treated with Peripheral scoring drug balloon.Dissolve AVF
  Interventions: Device: Dissolve AVF
- PTA Group (Active Comparator): This group treated with plain balloon catheter.Armada 35
  Interventions: Device: Armada 35

INTERVENTIONS:
Device: Dissolve AVF — Subjects in the test group will be treated with peripheral scoring drug balloon.
  Other Names: Using Peripheral scoring drug balloon catheter to cover the whole treated segment
  Arms: Dissolve AVF Group
Device: Armada 35 — Subjects in the test group will be treated with plain balloon catheter.
  Other Names: Using plain balloon catheter to cover the whole treated segment
  Arms: PTA Group

SUMMARY:
Drug-coated balloons delivering paclitaxel at the angioplasty site have proved their superiority in the treatment of coronary and peripheral arterial stenoses. Paclitaxel reduces neointimal hyperplasia, therefore, it represents an attractive option for AVF stenoses. This trial is aimed to evaluate the safety and efficacy of Peripheral scoring drug balloon (Dissolve AV) or Balloon Dilatation catheter ( Armada 35) in treating AVF stenosis in chinese population.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized controlled, open-label, superiority study. A total of 220 subjects will be enrolled from 11 sites in China. All subjects enrolled will be randomly assigned to the test group (Dissolve AV group, n=110) and the control group (Armada 35 group, n=110) with randomized allocation ratio of 1:1. Subjects in the test group and the control group will be treated with Peripheral scoring drug balloon or Balloon Dilatation catheter

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years (inclusive), male or female;
2. Patients with mature AVF/AVG and at least one successful hemodialysis session;
3. Target lesion located in the AVF/AVG reflux vein (excluding the feeding artery and central vein);
4. With hemodynamically significant AVF/AVG stenosis and meeting two of the following conditions (A & B) A. ≥ 50% stenosis of the target lesion as assessed by angiography B. Presence of at least one of the following (as defined in the NKF-K/DOQI guidelines) 1)Significantly elevated venous pressure during dialysis 2)Unexplained decrease in dialysis dose 3)Decrease in pump-controlled blood flow;
5. De novo or restenotic target lesion consisting of one or more tandem lesions, and with a visual reference vessel diameter of 4.0-8.0 mm and a total length ≤ 40 mm for the target lesion;
6. All non-target lesions must have <50% stenosis without clinical indication for treatment.
7. Patients who have signed the informed consent form.

Exclusion Criteria:

1. Patients who are participating in another clinical trial of a drug product or medical device;
2. Patients previously enrolled in this trial;
3. Women of childbearing age with a non-negative pregnancy test prior to surgical procedure, or lactating women;
4. Patients treated with major surgeries (e.g., open-heart surgery, cranial surgery) within 30 days prior to enrollment in the study;
5. Immature AVF/AVG (not subjected to dialysis; this vascular access has not been subjected to a single successful dialysis due to insufficient inner diameter that prevents successful puncture and results in inadequate blood flow);
6. Calcified lesions that are not expected to be dilated with a balloon;
7. AVF/AVG implanted with a stent;
8. AVF/AVG lesions previously treated with DCB;
9. Target lesions located at the venous anastomosis of AVF/AVG;
10. Impaired central venous reflux ;
11. Presence of a stenotic lesion in the artery that severely interferes with blood flow;
12. Patients with known allergy or intolerance to paclitaxel or contrast agent;
13. Patients with a life expectancy of less than 1 year;
14. Patients with concomitant systemic lupus erythematosus (SLE), ANCA-associated small vessel vasculitis;
15. Patients with a history of coagulopathy or thrombocytopenic purpura;
16. Patients treated with or scheduled to be treated with renal transplant or who have switched to peritoneal dialysis;
17. Vascular access infections or active systemic infections;
18. Presence of other medical conditions considered ineligible for the study as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2021-10-02 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Target lesion primary patency (TLPP) at 6 months post-procedure | 6 month post-procedure
  TLPP ends with postoperative target lesion (including 5 mm proximal and 5 mm distal to the target lesion) failure (TLF) or target lesion-associated vascular access thrombosis. TLF is defined as the presence of at least one clinical symptom of inadequate dialysis blood flow (as defined in the NKF-K/DOQI guidelines) due to stenosis of the target lesion (≥ 50% stenosis of the target lesion on imaging), including significantly elevated venous pressure during dialysis, abnormal physical examination findings, and a decrease in pump-controlled blood flow.

SECONDARY OUTCOMES:
Target lesion primary patency (TLPP) at 12 months post-procedure | 12 Month post-procedure
  TLPP ends with postoperative target lesion (including 5 mm proximal and 5 mm distal to the target lesion) failure (TLF) or target lesion-associated vascular access thrombosis. TLF is defined as the presence of at least one clinical symptom of inadequate dialysis blood flow (as defined in the NKF-K/DOQI guidelines) due to stenosis of the target lesion (≥ 50% stenosis of the target lesion on imaging), including significantly elevated venous pressure during dialysis, abnormal physical examination findings, and a decrease in pump-controlled blood flow.
Device success | 0 day post-procedure
  When evaluated with a single balloon dilatation catheter, it is defined as successful reach of a target lesion, dilatation without rupture, and successful withdrawal.
Procedural Success | 0 day post-procedure
  It is defined as ≤ 30% residual stenosis of the target lesion, and the absence of serious perioperative adverse events.
Clinical success | 0 - 5 days post-procedure
  At least one session of successful hemodialysis following the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: YE CHAOYANG, Study Chair — ShuGuang Hospital affiliated to Shanghai University of Traditional Chinese
Locations (10):
- China (10):
  - Emergency general hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Tongren hospital, Capital medical university, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - ShuGuang Hospital affiliated to Shanghai University of Traditional Chinese, Shanghai, Shanghai Municipality
  - Huashan hospital affiliated to FuDan university, Shanghai, Shanghai Municipality
  - Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Taiyuan Central Hospital, Taiyuan, Shanxi
  - Shaoyifu hospital, zhejiang medical universiyt, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No